CLINICAL TRIAL: NCT05280600
Title: Developing Advanced Neuroimaging for Clinical Evaluation of Autoimmune Encephalitis
Acronym: DANCE-AE
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Action Medical Research (Other)
Responsible Party: Sponsor
Other Study IDs: KCL21-018; GN2835 (Other Grant/Funding Number: Action Medical Research); IRAS 297793 (Other: Health Research Authority)
Record Dates: First submitted 2022-02-10; First posted 2022-03-15 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Autoimmune Encephalitis
Keywords: Magnetic resonance imaging (MRI); Magnetic resonance spectroscopy (MRS); Resting-state functional MRI; Cognition; Ultra-high field MRI
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NMDAR-antibody encephalitis: Children and young people (ages 8-24 years) with a diagnosis of NMDAR-antibody encephalitis.
  Interventions: Other: Not applicable - non-interventional study
- Antibody-negative autoimmune encephalitis: Children and young people (ages 8-24 years) with a diagnosis of autoantibody-negative but probable autoimmune encephalitis or definite autoimmune limbic encephalitis.
  Interventions: Other: Not applicable - non-interventional study
- Healthy control: Healthy children and young people (ages 8-24 years).
  Interventions: Other: Not applicable - non-interventional study

INTERVENTIONS:
Other: Not applicable - non-interventional study — Not applicable - non-interventional study

SUMMARY:
Autoimmune encephalitis is brain inflammation caused by the immune system mistakenly reacting against proteins in the brain. The commonest form is called NMDAR-antibody encephalitis (N-methyl-D-aspartate receptor antibody encephalitis), a rare condition which mainly affects children and young people and causes difficulties in memory, thinking and mental health which can have significant long-term impacts on education, employment and quality of life.

In this project we will use advanced magnetic resonance imaging (MRI) to measure changes in the structure, function and chemistry of the brains of children and young people who are in early recovery from NMDAR-antibody encephalitis and other forms of immune-mediated encephalitis. We will investigate if MRI measurements in patients differ from those in healthy people, and if they can help predict patient outcome one year later, assessed by tests of memory, thinking, mental health and functioning in daily life.

DETAILED DESCRIPTION:
This study aims to develop non-invasive, in vivo measures of neurobiological dysfunction derived from the overarching hypothesis that dysfunction of inhibitory interneurons alters the cerebral concentrations of gamma-aminobutyric acid (GABA) and glutamate (Glu) and underlies T2 changes and deficient connectivity in functional networks in early recovery from NMDAR-antibody encephalitis. Our ambition is to identify the best potential prognostic biomarkers from these neurometabolite measurements and structural and functional MRI.

Our primary objective is to test the following specific hypotheses in children and young people with NMDAR-antibody encephalitis:

* Hypothesis 1: GABA is decreased, and Glu increased, on MR spectroscopy of the medial temporal lobe and medial prefrontal cortex in NMDAR-antibody encephalitis.
* Hypothesis 2: Local GABA and Glu are correlated with (i) resting-state functional MRI (fMRI) based functional connectivity and (ii) parameter map-based microstructural changes. Specifically, we hypothesise that (i) GABA is positively correlated and Glu inversely correlated with functional connectivity, assessed by whole-brain mapping of the default mode network and seed-based analysis of hippocampal-frontal connectivity; and (ii) Glu is positively correlated and GABA inversely correlated with median T2 values within the hippocampus.
* Hypothesis 3: Local neurometabolites, network measures and microstructural changes predict cognitive, psychiatric and functional outcome at one year. Specifically, we hypothesise that medial temporal Glu, GABA and hippocampal T2 predict memory performance, and prefrontal Glu and GABA predict attention, executive function and fluid intelligence.

ELIGIBILITY:
INCLUSION CRITERIA:

NMDAR-antibody encephalitis group:

1. Age 8-24 years at study enrollment.
2. Disease onset in the last 12 months before study enrollment.
3. Meets consensus diagnostic criteria (Graus et al., 2016) for either probable anti-NMDAR encephalitis OR definite anti-NMDAR encephalitis.

Antibody-negative autoimmune encephalitis group:

1. Age 8-24 years at study enrollment.
2. Disease onset in the last 12 months before study enrollment.
3. Meets consensus diagnostic criteria (Graus et al., 2016) for either autoantibody-negative but probable autoimmune encephalitis OR definite autoimmune limbic encephalitis.

Healthy control group:

1. Age 8-24 years at study enrollment.

EXCLUSION CRITERIA:

All participants:

1. Any clear contra-indication for an MRI scan. In particular this would be due to the presence of any implanted devices or metal from previous surgery or accident.

Healthy control group:

1. A known neurological or neurodevelopmental disorder.

NMDAR-antibody encephalitis and antibody-negative autoimmune encephalitis groups:

1. Alternative more likely cause of neurological symptoms than autoimmune encephalitis, i.e. reasonable exclusion of other diagnoses as per consensus criteria (Graus et al., 2016).
2. Severe movement disorder/uncontrolled epilepsy/dysautonomia.
3. Previous infective encephalitis with major destructive brain lesions.

Ages: 8 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All participants will be recruited in the United Kingdom.
  NMDAR-antibody encephalitis and antibody-negative autoimmune encephalitis groups: Identified by neurologists/paediatric neurologists in secondary/tertiary healthcare settings, or by self-referral via the Encephalitis Society.
  Healthy control group: Identified from King's College London volunteer databases, friends and siblings of autoimmune encephalitis cases, or recruited from local schools and colleges.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Cerebral concentrations of GABA and glutamate at the prefrontal cortex and left medial temporal lobe | Baseline
  Measured with MR spectroscopy - stimulated echo acquisition mode (STEAM) sequence
Structural MRI | Baseline
  Quantitative MRI parameter maps including measurement of median T2 values in the hippocampus
Resting-state fMRI | Baseline
  Whole-brain mapping of the default mode network and seed-based analysis of hippocampal-frontal connectivity

SECONDARY OUTCOMES:
Wechsler Abbreviated Scale of Intelligence 2nd Edition (WASI-II) | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
Rey Auditory Verbal Learning Test (RAVLT) | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
Doors & People Test | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
CANTAB (Cambridge Cognition, UK): Paired Associates Learning | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
CANTAB (Cambridge Cognition, UK): Rapid Visual Information Processing | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
CANTAB (Cambridge Cognition, UK): Spatial Span | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
CANTAB (Cambridge Cognition, UK): Intra-Extra Dimensional Set Shift | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
CANTAB (Cambridge Cognition, UK): Stockings of Cambridge | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
CANTAB (Cambridge Cognition, UK): Stop Signal Task | Baseline (all groups), 1 year (patients)
  Cognitive test (higher score indicating better outcome)
Prodromal Questionnaire Brief Version (PQ-B) | Baseline (all groups), 1 year (patients)
  Questionnaire-based psychiatric symptom score (lower score indicating better outcome)
Patient Health Questionnaire (PHQ-9) | Baseline (all groups), 1 year (patients)
  Questionnaire-based psychiatric symptom score (lower score indicating better outcome)
Generalized Anxiety Disorder 7-item Scale (GAD-7) | Baseline (all groups), 1 year (patients)
  Questionnaire-based psychiatric symptom score (lower score indicating better outcome)
Pediatric Quality of Life Inventory (PedsQL) Generic Core Scales | Baseline (all groups), 1 year (patients)
  Questionnaire-based functional outcome score (higher score indicating better outcome)
PedsQL Multidimensional Fatigue Scale | Baseline (all groups), 1 year (patients)
  Questionnaire-based functional outcome score (higher score indicating better outcome)
Behaviour Rating Inventory of Executive Function (BRIEF) | Baseline (all groups), 1 year (patients)
  Questionnaire-based functional outcome score (lower score indicating better outcome)
Conners 3 Short Form / Conners' Adult ADHD Rating Scale | Baseline (all groups), 1 year (patients)
  Questionnaire-based functional outcome score (lower score indicating better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: David W Carmichael, PhD MSci, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Consent will be requested from participants to share imaging data and summary clinical and demographic data. Where participants consent, imaging data will be de-identified, removing facial features from the magnetic resonance images and all identifying information will be removed from the image header (the part of the file that describes how the image data was acquired). The resulting data will be shared together with anonymised clinical data at the request of other researchers.
Time Frame: To be confirmed
Access Criteria: Requests for data access from researchers at accredited research institutions will be considered. Any requests for data sharing may require a formal agreement to be put in place between the Sponsors and the recipient.

REFERENCES:
- [Background] Graus F, Titulaer MJ, Balu R, Benseler S, Bien CG, Cellucci T, Cortese I, Dale RC, Gelfand JM, Geschwind M, Glaser CA, Honnorat J, Hoftberger R, Iizuka T, Irani SR, Lancaster E, Leypoldt F, Pruss H, Rae-Grant A, Reindl M, Rosenfeld MR, Rostasy K, Saiz A, Venkatesan A, Vincent A, Wandinger KP, Waters P, Dalmau J. A clinical approach to diagnosis of autoimmune encephalitis. Lancet Neurol. 2016 Apr;15(4):391-404. doi: 10.1016/S1474-4422(15)00401-9. Epub 2016 Feb 20. PMID 26906964